CLINICAL TRIAL: NCT02792543
Title: Impact of Chyme Reinfusion Compared to Parenteral Nutrition on the Incidence of Complications in Patients With a Temporary High-output Double Enterostomy: a Multicentre Randomized Controlled Trial - FRY: efFiciency of Reinfusion of chYme - (FRY)
Acronym: FRY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL16_0098
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Intestinal Failure With a Temporary High-output Double Enterostomy
Keywords: nutrition; double enterostomy; chyme reinfusion; randomized controlled trial
MeSH Terms: interventions — Parenteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- parenteral nutrition (Active Comparator): Parenteral nutrition consists of electrolyte supplementation, hydration, and nutrition through a central venous catheter.
  Interventions: Drug: parenteral nutrition
- chyme reinfusion (Experimental): Chyme reinfusion consists of continuously reinfusing the chyme collected from the proximal small bowel segment via the enterostomy, and into the diverted distal small bowel segment. It implies the use of the Entéromate™ pump.
  Interventions: Device: Entéromate™

INTERVENTIONS:
Device: Entéromate™ — Chyme reinfusion (the experimental treatment) consists of continuously reinfusing the chyme collected from the proximal small bowel segment via the enterostomy, and into the diverted distal small bowel segment. It implies the use of the Entéromate™ pump.
  Other Names: chyme reinfusion
  Arms: chyme reinfusion
Drug: parenteral nutrition — Parenteral nutrition (the gold standard treatment) consists of electrolyte supplementation, hydration, and nutrition through a central venous catheter.
  Arms: parenteral nutrition

SUMMARY:
In the case of intestinal failure with a high-output double enterostomy, the parenteral nutrition (PN) is the gold standard treatment until the surgical reestablishment of digestive continuity. PN has its own morbidity, and in the absence of expertise, the risks of infectious, mechanical, and metabolic complications are increased. Chyme reinfusion (CR) is an enteral nutritional technique which reestablishes the functional continuity of the anatomically present small bowel through an extracorporeal circulation of the chyme. In patients with intestinal failure with a temporary high-output double enterostomy, we hypothesize that CR, compared to PN will reduce post-operative complications after surgical reestablishment of digestive continuity, maintain the intestinal function including absorption, and reduce the complications during the transitional period pending the surgical reestablishment of digestive continuity.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Temporary high-output double enterostomy (≥1500ml/24 hours)
* Total small bowel length ≥ 120 cm
* Downstream small bowel consisting of at least 25 cm of healthy bowel, accessible by a stoma, and suitable for chyme reinfusion
* Oral feeding resumed for at least 5 days
* Parenteral nutrition or hydration required until the surgical reestablishment of digestive continuity
* Affiliation to an health insurance (general Social Security scheme or an equivalent scheme)
* No current or planned participation in another biomedical research
* Signature of an informed consent form

Exclusion Criteria:

* Expected duration of parenteral nutrition or chyme reinfusion less than 2 weeks
* Refusal by the patient to have a mixed texture diet,
* Chemotherapy or radiotherapy before the surgical reestablishment of digestive continuity,
* Not drained intra-abdominal collection,
* Fever, uncontrolled infection, or infection treated for less than 72 hours,
* Shock of any cause,
* Creatinine clearance ≤ 60 ml/min
* Patients under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
The frequency of complications occurring in patients with a temporary high-output double enterostomy. | From the day which the patient no longer requires surgical care after the surgical placement of a temporary double enterostomy (Day 0) and up to 30 days after the reestablishment of digestive continuity (Month 4 (minus) - Month 9 (plus))
  The reestablishment of digestive continuity is possible between Month 3 and Month 8 (it is patient-dependent) The complications, and their severity, will be classed using the Dindo-Clavien classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital de la Croix Rousse, Lyon, France